CLINICAL TRIAL: NCT03425474
Title: A Phase Ⅲ, Multicentre, Randomized, Single-blinded Study to Evaluate the Safety and Efficacy of the Sedation for Remimazolam or Propofol in Patients Undergoing Diagnostic Upper GI Endoscopy
Brief Title: Study of Remimazolam Tosilate in Patients Undergoing Diagnostic Upper GI Endoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HR-RMZL-Ⅲ-UGE
Record Dates: First submitted 2017-09-16; First posted 2018-02-07 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Tosilate (Experimental): Remimazolam Tosilate at 5mg for initial dose
  Interventions: Drug: Remimazolam Tosilate
- Propofol (Active Comparator): Propofol at 1.5mg/kg for initial dose
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam Tosilate — Initial dose plus supplemental doses as necessary
  Arms: Remimazolam Tosilate
Drug: Propofol — Initial dose plus supplemental doses as necessary
  Arms: Propofol

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the sedation for Remimazolam or Propofol in patients undergoing diagnostic upper GI endoscopy.

DETAILED DESCRIPTION:
This is a multi-center, ,parallel-group, single blind study using Remimazolam or propofol for sedation in patients undergoing diagnostic upper GI endoscopy.Subjects are randomized to different treatment groups (including 1 for Remimazolam Tosilate and 1 for propofol). Fentanyl are permitted during a diagnostic upper GI endoscopy.Efficacy and safety profiles of Remimazolam Tosilate are to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 18-60 years；
* intending to undergo diagnostic upper GI endoscopy;
* ASA( American Society of Anesthesiologists) I or II；
* 18 kg/m²<BMI(Body Mass Index)<30 kg/m²;
* the operation time of gastroscopy is not more than 30 min；
* Signed informed consent.

Exclusion Criteria:

* Patients need to be Complicated gastroscopy;
* Patients need to be Tracheal intubation;
* Patients with respiratory management difficulties (Modified Mallampati grade IV）;
* one or more of the laboratory findings fall out of the limitations for this study(platelet,hemoglobin,aspartate aminotransferase,etc.);
* A history of drug abuse and / or alcohol abuse 2 years prior to the screening period；
* allergic to drugs used in the study;
* pregnant women or those in lactation period
* The subject has participated in other clinical trial within the 3 months prior to randomization.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 378 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
rate of successful sedation | approximately 3 hours
  successful sedation rate as measured by the proportion of subjects who experienced successful sedation during diagnostic upper GI endoscopy.

SECONDARY OUTCOMES:
Sedation induction time | approximately 3 hours
  Sedation induction time is defined as from start of study drug injection to the first time of MOAA/S（The Observer's Assessment of Alertness/Sedation Scale） ≤ 3.
Sedation recovery time | approximately 3 hours
  Sedation induction time is defined as from stop of study drug injection to be wide awake.
rate of hypotension | approximately 3 hours
  rate of hypotension as measured by the proportion of subjects who experienced hypotension during a diagnostic upper GI endoscopy
rate of respiratory depression | approximately 3 hours
  rate of respiratory depression as measured by the proportion of subjects who experienced respiratory depression during a diagnostic upper GI endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical trial Ethnics Committee of Peking Union Medical College Hospital, Beijing, Beijing Municipality, China